CLINICAL TRIAL: NCT04537546
Title: EVINOV: Prevention of Abdominal Incisional Hernia After Laparoscopic Digestive Surgery in Obese Patients (BMI>30kg/m2)
Brief Title: Prevention of Abdominal Incisional Hernia After Laparoscopic Digestive Surgery in Obese Patients (BMI>30kg/m2)
Acronym: EVINOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DIG-02-2018
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: Laparoscopy; Eventration; Abdominal support belt
MeSH Terms: conditions — Obesity; Gastroschisis

STUDY DESIGN:
Intervention Model Description: Feasibility study, single arm, interventional and prospective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elasto compression belt (Experimental): all patients must wear the belt 2 months after laparoscopic digestive surgery.
  Interventions: Device: OBESINOV elasto-compressive belt

INTERVENTIONS:
Device: OBESINOV elasto-compressive belt — It is a customised medical device, using a technique for calculating the compression ratio adapted to each patient according to his morphology

SUMMARY:
The hypothesis of this study is to show that after laparoscopic digestive surgery in obese patients (BMI>30kg/m2), the wearing of an abdominal support belt is an effective treatment for the Incisional Hernia and feasible in terms of compliance, quality of life and patient satisfaction

DETAILED DESCRIPTION:
The study will be conducted at the Institut Mutualiste Montsouris, it is planned to include 350 patients in 12 months, the duration of participation of each patient is 24 months.

An orthopaedist will see patients in consultation to take their measurements, patients complete a quality of life questionnaire (the SF 36), when they are admitted for surgery.

After surgery, patients begin wearing their belts according to the instructions given by the surgeon during hospitalization:

* Start wearing the belt as soon as possible.
* wear it according to its recommendations: all day, every day of the week and for two months.

Patients should record the number of hours they would have worn their belts in the EVINOV logbook each day.

The studu Co will contact patients by phone every two weeks for the 2 months they will be wearing the belt.

At the one-month post-operative consultation, the patient will complete a quality of life questionnaire again (the SF 36).

Two months after surgery, patients receive a final SF 36 questionnaire by mail, with a satisfaction scale to evaluate their overall feeling around the period of wearing the abdominal belt. Patients are asked to return these two documents, as well as the EVINOV logbook.

The latest health data collection is the imaging data from the abdominal CT scan at 24 months, which will show the presence or absence of an incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 years of age.
* Signed an informed consent form (ICF) indicating that the subject understands the purpose of and procedures required for the study.
* Having a BMI >30kg/m2.
* Affiliated to health insurance regimen.
* Having undergone laparoscopic digestive surgery

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Patient under guardianship or unable to give consent.
* People particularly protected by French law.
* Having undergone laparoscopic digestive surgery with ileostomy or ostomy closure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Presence or not of an eventration | During the 24 months following sugery
  The presence of the eventration is detected by an abdominal CT scan.

SECONDARY OUTCOMES:
Patient satisfaction: 5 level Likert scale2 | 2 months after surgery
  The satisfaction of patient is evaluated by the 5 level Likert scale2
Quality of life of patients: SF-36 quetionnaire | before surgery, 1 month after surgery and 2 months after surgery.
  The quality of life of patients is evaluated using SF-36 quetionnaire.
Compliance with preventive treatment by the abdominal support belt. | 2 months after surgery
  Patient compliance collected through a logbook completed daily.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pourcher, Dr, Study Chair — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Lee DY, Rehmani SS, Guend H, Park K, Ross RE, Alkhalifa M, McGinty JJ, Teixeira JA. The incidence of trocar-site hernia in minimally invasive bariatric surgery: a comparison of multi versus single-port laparoscopy. Surg Endosc. 2013 Apr;27(4):1287-91. doi: 10.1007/s00464-012-2597-5. Epub 2012 Dec 12. PMID 23232997
- [Background] Agaba EA, Rainville H, Ikedilo O, Vemulapali P. Incidence of port-site incisional hernia after single-incision laparoscopic surgery. JSLS. 2014 Apr-Jun;18(2):204-10. doi: 10.4293/108680813X13693422518317. PMID 24960483
- [Background] Bosanquet DC, Ansell J, Abdelrahman T, Cornish J, Harries R, Stimpson A, Davies L, Glasbey JC, Frewer KA, Frewer NC, Russell D, Russell I, Torkington J. Systematic Review and Meta-Regression of Factors Affecting Midline Incisional Hernia Rates: Analysis of 14,618 Patients. PLoS One. 2015 Sep 21;10(9):e0138745. doi: 10.1371/journal.pone.0138745. eCollection 2015. PMID 26389785
- [Background] Weissler JM, Lanni MA, Hsu JY, Tecce MG, Carney MJ, Kelz RR, Fox JP, Fischer JP. Development of a Clinically Actionable Incisional Hernia Risk Model after Colectomy Using the Healthcare Cost and Utilization Project. J Am Coll Surg. 2017 Aug;225(2):274-284.e1. doi: 10.1016/j.jamcollsurg.2017.04.007. Epub 2017 Apr 23. PMID 28445797